CLINICAL TRIAL: NCT05309421
Title: An Open Label, Single Arm Trial Evaluating the Efficacy and Safety of EVX-01 in Combination With Pembrolizumab in Checkpoint Inhibitor Treatment naïve Adults With Unresectable or Metastatic Melanoma
Brief Title: A Single Arm Trial Evaluating the Efficacy and Safety of EVX-01 in Combination With Pembrolizumab in Adults With Unresectable or Metastatic Melanoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Evaxion Biotech A/S (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EVX-01-001; 2024-512393-10-00 (EU CTIS Number); KEYNOTE-D36 (Other: Merck Sharp & Dohme Corp.)
Record Dates: First submitted 2022-03-22; First posted 2022-04-04 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Melanoma Stage IV; Unresectable Melanoma
Keywords: Personalized immunotherapy; Personal cancer vaccine; cancer vaccine; EVX-01
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- EVX-01 in combination with pembrolizumab (Experimental): EVX-01 is administered im. Pembrolizumab is administered according to label
  Interventions: Drug: EVX-01; Drug: Pembrolizumab 25 MG/ML

INTERVENTIONS:
Drug: EVX-01 — Investigational drug given in combination with standard of care
Drug: Pembrolizumab 25 MG/ML — Standard of care
  Other Names: Keytruda

SUMMARY:
The purpose of this single arm, multi-national clinical trial in patients with metastatic or unresectable melanoma is to evaluate the BOR and compare it to historical data on patients on anti-PD1 treatment with pembrolizumab alone.

DETAILED DESCRIPTION:
Patients will initiate treatment with pembrolizumab at the start of the trial and receive up to 18 treatment cycles (approximately 2 years). Immunization with the EVX-01 will be initiated at Week 12. In total, 10 doses of EVX-01 will be administered intramuscularly, with 6 doses given two weeks apart and 4 booster doses at later time points.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age on day of signing informed consent.
* Histologically confirmed, and not amenable to local therapy, metastatic or unresectable melanoma Stage III or Stage IV, as per AJCC 8th ed. staging system.

  1. Patient may not have a diagnosis of uveal or ocular melanoma.
  2. Patients must be treatment naïve to checkpoint inhibitor (CPI) therapy
  3. Patients must have testing for a BRAF mutation prior to study entry.

Note: Patients with BRAF V600E mutant melanoma may have received prior BRAF inhibitor therapy as first-line systemic therapy and be eligible for this study as second line treatment. At the discretion of the investigator, patients with BRAF V600E mutant melanoma who have NOT received a BRAF inhibitor are also eligible for this study as first line treatment if they meet the following additional criteria:

i. LDH < local ULN, ii. No clinically significant tumor related symptoms in the judgment of the investigator, and iii. Absence of rapidly progressing metastatic melanoma in the judgment of the investigator

* Have measurable disease per RECIST 1.1 as assessed by the local site investigator within 4 weeks prior to the first visit. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* Patients must be willing and able to provide fresh or frozen tumor tissue from an unresectable or metastatic site of disease for neoepitope and biomarker analyses. If a sufficient amount of tumor tissue from an unresectable or metastatic site is not available prior to the start of the screening phase, subjects must consent to allow the acquisition of additional tumor tissue. In addition, participants may provide additional biopsy at the time of discontinuation due to progression.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

Exclusion Criteria:

* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137).
* Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to treatment.
* Has received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
* Has received a live or live-attenuated vaccine within 30 days prior to the first dose of study intervention. Note: Administration of killed vaccines are allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Change in the best overall response (BOR) | Measurements at Baseline through study completion (up to 102 weeks)
  Composite of a BOR of complete response (CR) or PR for patients with SD at the time of first EVX-01 administration and a BOR of CR for patients with PR at the time of first EVX-01 administration, within 2 years of treatment with pembrolizumab, as per RECIST 1.1 criteria

SECONDARY OUTCOMES:
Change in overall response rate | Measurements at Baseline through study completion (up to 102 weeks)
  Overall response rate, defined as the proportion of the patients who have best response as CR or PR assessed 2 years after initiation of treatment with pembrolizumab, as per RECIST 1.1 criteria
Change in progression free survival (PFS) | Measurements at Baseline through study completion (up to 102 weeks)
  PFS in patients with an assessment of SD, PR, or CR at the time of first EVX-01 administration, assessed 2 years after initiation of treatment with pembrolizumab and defined as the time from the first EVX-01 administration to the first documented disease progression per RECIST 1.1. criteria or death due to any causes, whichever occurs first
Change in overall survival (OS) | Measurements at Baseline through study completion (up to 102 weeks)
  OS assessed 2 years after initiation of treatment with pembrolizumab and defined as the time from initiation of treatment of pembrolizumab to death due to any cause
Number, type and severity of adverse events (AEs) and serious adverse events (SAEs) | Measurements at Baseline through study completion (up to 102 weeks)
  Number, type and severity of adverse events (AEs) and serious adverse events (SAEs)
Immunologic response induced by EVX-01 | Measurements at Baseline through study completion (up to 102 weeks)
  Activation and level of neoepitope specific T-cells before, during and after EVX-01 immunization
Percentage of patients in which EVX-01 is generated, produced, and administered | From tumor biopsy sampling to first dose of EVX-01 (up to 16 weeks)
  Percentage of patients in which EVX-01 is generated, produced, and administered

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (2):
  - Melanoma Institute Australia, Wollstonecraft, New South Wales
  - One Clinical Research, Nedlands, Western Australia
- Italy (2):
  - Divisione di Oncologia Medica del Melanoma, Milan
  - Instituto Nazionale Tumori IRCCS Fondazione, Napoli

REFERENCES:
- [Derived] Long GV, Ferrucci PF, Khattak A, Meniawy TM, Ott PA, Chisamore M, Trolle T, Hyseni A, Heegaard E. KEYNOTE - D36: personalized immunotherapy with a neoepitope vaccine, EVX-01 and pembrolizumab in advanced melanoma. Future Oncol. 2022 Oct;18(31):3473-3480. doi: 10.2217/fon-2022-0694. Epub 2022 Sep 1. PMID 36047545
- See also: PR — https://investors.evaxion.ai/node/9851/pdf